CLINICAL TRIAL: NCT06987448
Title: Clinical Comparison of CAD/CAM Nanohybrid Composite and Hybrid Ceramic Overlays in Children With Molar-Incisor Hypomineralisation: a Split-mouth Prospective Randomized Clinical Trial
Brief Title: Clinical Comparison of CAD/CAM Nanohybrid Composite and Hybrid Ceramic Overlays in Children With Molar-Incisor Hypomineralisation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alp Akça (Other)
Collaborators: Marmara University (Other)
Responsible Party: Sponsor-Investigator, Alp Akça, Principal Investigator, Marmara University
Organization: Marmara University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MUPEDDENTALPAKCA
Record Dates: First submitted 2025-05-07; First posted 2025-05-23 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Enamel Hypoplasia; Molar-Incisor Hypomineralization (MIH); Restoration of Permanent Molars Affected by MIH With CAD/CAM Blocks
Keywords: Molar-Incisor Hypomineralization; Pediatric Dentistry; Digital Workflow; Tooth Sensitivity; Immediate Dentin Sealing
MeSH Terms: conditions — Dental Enamel Hypoplasia; Molar Hypomineralization; Dentin Sensitivity

STUDY DESIGN:
Intervention Model Description: The study involves the application of a hybrid composite CAD/CAM restoration to one of two permanent first molar teeth affected by MIH in each patient, and a hybrid ceramic CAD/CAM restoration to the other tooth.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hybrid Composite Block Group (HCB) (Experimental): In this group, semi-direct onlay restorations were applied using nano-ceramic hybrid composite blocks (Grandio blocs, VOCO) fabricated through a CAD/CAM digital workflow. Following cavity preparation, dentin surfaces were sealed using the Immediate Dentin Sealing (IDS) technique. The restorations were cemented with a dual-cure resin cement
  Interventions: Procedure: Semi-direct onlay restoration using CAD/CAM hybrid ceramic block
- Hybrid Ceramic Block Group (HCB) (Experimental): In this group, onlay restorations were fabricated from polymer-infiltrated feldspathic ceramic blocks (VITA Enamic) using a CAD/CAM-assisted digital workflow. After hydrofluoric acid etching and silane application to the internal surface of the restoration, IDS-treated tooth surfaces were prepared for cementation. Restorations were bonded using a dual-cure resin cement.
  Interventions: Procedure: Semi-direct onlay restoration using CAD/CAM hybrid composite block

INTERVENTIONS:
Procedure: Semi-direct onlay restoration using CAD/CAM hybrid composite block — This refers to restorations fabricated from nano-ceramic hybrid composite blocks via chairside CAD/CAM workflow and cemented to permanent molars affected by MIH (molar-incisor hypomineralization).
  Arms: Hybrid Ceramic Block Group (HCB)
Procedure: Semi-direct onlay restoration using CAD/CAM hybrid ceramic block — This refers to restorations fabricated from polymer-infiltrated hybrid ceramic blocks using a digital workflow, then cemented to MIH-affected permanent molars.
  Arms: Hybrid Composite Block Group (HCB)

SUMMARY:
This clinical study was conducted to compare two different dental materials used in the treatment of children who have a condition called molar-incisor hypomineralization (MIH). MIH affects the quality of the enamel in permanent molars and can cause sensitivity, pain, and rapid tooth breakdown. In this study, children between the ages of 8 and 13 who had MIH in at least two molars received two types of onlay restorations: one made from a hybrid composite block and the other from a hybrid ceramic block. Both restorations were designed and manufactured using a digital system called CAD/CAM, which allows for more precise and efficient dental treatment.

Each child received both types of restorations-one on each side of the mouth-in a split-mouth design. The goal was to see how well each material worked over a period of six months. The restorations were evaluated by trained dentists using clinical criteria, and the children were also assessed for tooth sensitivity using a cold air test.

The main purpose of this study was to find out which material provides better clinical performance and reduces tooth sensitivity more effectively.

DETAILED DESCRIPTION:
Molar-Incisor Hypomineralization (MIH) is a developmental enamel defect that primarily affects the first permanent molars and frequently the incisors. It is characterized by hypomineralized enamel with increased porosity, discoloration, and a high risk of post-eruptive enamel breakdown. Affected teeth often present with significant sensitivity, posing difficulties in achieving adequate anesthesia and effective bonding during restorative procedures. As a result, the management of MIH-affected molars in pediatric patients is both complex and clinically significant.

This prospective, randomized, split-mouth clinical study was designed to compare two different CAD/CAM materials used in semi-direct onlay restorations for the treatment of MIH-affected molars in children aged 8 to 13 years. The materials under investigation were a nano-hybrid composite block (Grandio blocs, VOCO) and a polymer-infiltrated ceramic network (PICN) hybrid ceramic block (VITA Enamic, VITA Zahnfabrik).

The study enrolled 20 pediatric patients, each presenting with at least two permanent first molars affected by MIH (classified as score 2b/c or 4b/c according to the MIH-TNI criteria). Using a split-mouth design, each patient received both interventions-one molar restored with a hybrid composite block and the other with a hybrid ceramic block. Randomization was performed using a computer-generated sequence. All procedures were carried out by a trained pediatric dentistry resident under rubber dam isolation, following a standardized adhesive protocol.

The restorative process was completed in a single session and followed a fully digital workflow. Teeth were scanned intraorally using the CEREC system, and restorations were designed and milled chairside. Immediate dentin sealing (IDS) was applied prior to cementation. The internal surfaces of the restorations were prepared using appropriate surface treatments such as sandblasting or hydrofluoric acid etching followed by silane application, in accordance with the manufacturers' guidelines. Final cementation was performed using a dual-cure resin cement.

Follow-up evaluations are planned at 6, 12, and 18 months post-operatively. At each time point, clinical assessments are conducted by two calibrated, blinded evaluators using modified United States Public Health Service (USPHS) criteria. These include evaluations of marginal adaptation, surface integrity, anatomical form, marginal discoloration, and the presence of secondary caries. Additionally, thermal sensitivity is assessed using the Schiff Cold Air Sensitivity Scale to monitor changes in dentin hypersensitivity over time.

This study aims to provide comparative data on the mid-term clinical performance of two innovative restorative materials applied in MIH-affected molars using a minimally invasive, digital workflow.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 8 and 13 years
* Presence of at least two permanent first molars affected by MIH
* MIH-affected molars classified as score 2b, 2c, 4b, or 4c according to the MIH-TNI index
* Symmetrical molars suitable for split-mouth comparison
* Cooperative behavior sufficient to allow treatment under local anesthesia
* Signed informed consent obtained from parent or legal guardian

Exclusion Criteria:

* Presence of systemic or syndromic diseases affecting enamel development
* History of bruxism or parafunctional habits
* Presence of pulp involvement, fistula, or periapical pathology in the target teeth
* Allergies to dental materials used in the study (e.g., resin-based composites, adhesives)
* Participation in another clinical trial within the past 30 days
* Inability to attend scheduled follow-up appointments at 6, 12, and 18 months

Use of medication affecting pain perception or healing process

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2023-09-11 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2025-09-11 (Actual)

PRIMARY OUTCOMES:
Clinical performance of onlay restorations based on modified USPHS criteria | 6, 12, and 18 months post-treatment
  Assessment of the clinical acceptability of CAD/CAM-fabricated semi-direct onlay restorations using modified United States Public Health Service (USPHS) criteria, including Surface luster/roughness, Surface and marginal staining, Color match, Anatomic form, Fracture of restoration, Marginal adaptation, Patient's view, Postop. hypersensitivity and tooth vitality, Recurrence of erosion/caries and Fracture of tooth
  Scores:
  Acceptable:
  1. Perfect
  2. Good
  3. Acceptable
     Unacceptable (failed):
  4. Bad
  5. Gross

SECONDARY OUTCOMES:
Dentin hypersensitivity assessed by the Schiff Cold Air Sensitivity Scale | Baseline (pre-treatment), 6 months, 12 months, and 18 months post-treatment
  Evaluation of thermal sensitivity in restored MIH-affected molars using the Schiff Cold Air Sensitivity Scale. The test involves applying a standardized air stimulus to the tooth surface and scoring the response on a scale from 0 to 3. Ordinal (Schiff scale: 0 = no response, 1 = response but no request to stop, 2 = response with request to stop, 3 = painful response)
Intra-examiner and inter-examiner agreement on clinical evaluation criteria | At each clinical follow-up visit (6, 12, and 18 months)
  Measurement of the consistency and reliability between two calibrated evaluators in assessing clinical performance using modified USPHS criteria. Agreement will be calculated using kappa statistics. Statistical agreement (Cohen's Kappa coefficient) Assessment of the clinical acceptability of CAD/CAM-fabricated semi-direct onlay restorations using modified United States Public Health Service (USPHS) criteria, including Surface luster/roughness, Surface and marginal staining, Color match, Anatomic form, Fracture of restoration, Marginal adaptation, Patient's view, Postop. hypersensitivity and tooth vitality, Recurrence of erosion/caries and Fracture of tooth
  Scores:
  Acceptable:
  1. Perfect
  2. Good
  3. Acceptable
     Unacceptable (failed):
  4. Bad
  5. Gross

CONTACTS AND LOCATIONS:
Overall Officials: Alp Akça, Doctor of Dental Surgery (DDS), Principal Investigator — Marmara University, School of Dentistry, Department of Pediatric Dentistry
Locations (1):
- Marmara University, School of Dentistry, Department of Pediatric Dentistry. Marmara Üniversitesi Sağlık Yerleşkesi, Diş Hekimliği Fakültesi, Başıbüyük Yolu 9/3 34854 Başıbüyük / Maltepe / İSTANBUL., Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (including intraoral photographs and clinical evaluation scores) may be shared in scientific publications or presentations. Data will be limited to information relevant for scientific analysis and will not include any personal identifiers.
Supporting Information: Study Protocol, SAP
Time Frame: De-identified individual participant data (IPD), along with supporting documents such as the study protocol and statistical analysis plan, will be available beginning 6 months after publication of the primary study results and will remain available for 5 years following the publication date.
Access Criteria: Requests for access to de-identified individual participant data and supporting documents will be considered for academic or scientific research purposes. Interested researchers must submit a written proposal detailing the planned analysis, including objectives and statistical methods. Requests will be reviewed by the principal investigator and institutional review board (IRB) representatives to ensure ethical compliance and scientific merit. A data use agreement must be signed prior to data release. Requests can be submitted via email to the corresponding author listed in the publication.